CLINICAL TRIAL: NCT07377981
Title: An Exploratory Study of the Efficacy and Safety of Esketamine and Dexmedetomidine in Non-Intubated ICU Patients With Hyperactive Delirium
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-SR-1088
Record Dates: First submitted 2026-01-12; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Dexmedetomidine; Ketamine; Analgesia; Respiratory Therapy; Intensive Care Units (ICUs); Agitation; Sedation and Analgesia
Keywords: Sedation and analgesia; Analgesia; Agitation; Dexmedetomidine; Ketamine; Intensive Care Units (ICUs); Respiratory Therapy
MeSH Terms: conditions — Agnosia; Psychomotor Agitation | interventions — Dexmedetomidine; Fumigant 93

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine combined with dexmedetomidine (Experimental): Patients will receive a loading dose of esketamine at 0.1 mg/kg (subanesthetic dose) without a concomitant loading dose of dexmedetomidine. This will be followed by a continuous intravenous infusion (pump-driven) of esketamine at 0.125-0.20 mg/(kg·h) (subanesthetic dose) combined with dexmedetomidine at 0.2-0.5 μg/kg/h. The infusion will be maintained until the patient fulfills the criteria of both a negative CAM-ICU assessment and a RASS score between -2 and +1.
  Interventions: Drug: Esketamine combined with dexmedetomidine
- Dexmedetomidine (Active Comparator): Patients will receive a loading dose of normal saline (0.1 mL/kg), without a loading dose of dexmedetomidine. This will be followed by a continuous intravenous infusion (pump-driven) of normal saline at an equivalent volume to the esketamine infusion rate (simulating 0.125-0.20 mg/(kg·h)), combined with dexmedetomidine at 0.2-0.5 μg/kg/h. The infusion will be continued until the patient meets both criteria: a negative CAM-ICU assessment and a RASS score between -2 and +1.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Esketamine combined with dexmedetomidine — Patients will receive a loading dose of esketamine at 0.1 mg/kg (subanesthetic dose) without a concomitant loading dose of dexmedetomidine. This will be followed by a continuous intravenous infusion (pump driven) of esketamine at 0.125-0.20 mg/(kg·h) (subanesthetic dose) combined with dexmedetomidine at 0.2-0.5 μg/kg/h. The infusion will be maintained until the patient fulfills the criteria of both a negative CAM ICU assessment and a RASS score between -2 and +1.
  Other Names: E+D
  Arms: Esketamine combined with dexmedetomidine
Drug: Dexmedetomidine — Patients will receive a loading dose of normal saline (0.1 mL/kg), without a loading dose of dexmedetomidine. This will be followed by a continuous intravenous infusion (pump driven) of normal saline at an equivalent volume to the esketamine infusion rate (simulating 0.125-0.20 mg/(kg·h)), combined with dexmedetomidine at 0.2-0.5 μg/kg/h. The infusion will be continued until the patient meets both criteria: a negative CAM ICU assessment and a RASS score between -2 and +1.
  Other Names: D
  Arms: Dexmedetomidine

SUMMARY:
This investigator-initiated, randomized, controlled, superiority trial aims to assess the efficacy and safety of esketamine combined with dexmedetomidine for the management of agitation or delirium in intensive care unit (ICU) patients receiving non-invasive respiratory support. The primary endpoint is the duration of delirium.

DETAILED DESCRIPTION:
Delirium is defined as an acute disturbance in attention and consciousness that develops over a short period of time and is accompanied by other cognitive impairments, such as memory deficits, disorientation, or perceptual abnormalities. It represents the most common clinical manifestation of acute brain dysfunction in the intensive care unit (ICU). Based on psychomotor activity, delirium is classified into three subtypes: hyperactive, hypoactive, and mixed. Hyperactive delirium is the most readily recognized form, characterized by agitation, emotional lability, hallucinations, or delusions. Patients with this subtype often exhibit impulsive behaviors-such as attempting to remove intravenous lines in the ICU-which can lead to serious injury or life-threatening situations. Furthermore, agitation induces a state of physiological stress, amplifies neuroendocrine responses, increases organ load, and may exacerbate the underlying illness. For instance, it can elevate blood pressure, raise heart rate, and increase oxygen consumption, potentially triggering cardiac or cerebrovascular events in patients with preexisting conditions. During episodes of agitation or delirium, inflammatory markers such as IL 6, IL 8, IL 2, and CRP are elevated. The rise in pro inflammatory cytokines activates microglia, leading to further release of inflammatory mediators and creating a vicious cycle that exacerbates neuroinflammation. According to the Chinese Guidelines for Pain and Sedation in Adult ICU Patients, delirium is a risk factor for poor prognosis in ICU patients, not only increasing mortality and extending hospital stay but also imposing a significant economic burden. Given these adverse consequences, the early management of delirium in the ICU is particularly important.

Treatment strategies for delirium include non pharmacological approaches, such as those incorporated into bundled care models like the ABCDE bundle, which have been shown to support recovery. While the ABCDE bundle is supported by high quality evidence regarding its efficacy and safety, its complexity often makes full implementation challenging in clinical practice, leading to greater reliance on pharmacological interventions. Pharmacological prevention may include supplements such as melatonin to improve sleep quality and avoid sleep deprivation associated delirium. The selective melatonin receptor agonist ramelteon shortens sleep latency and promotes sleep maintenance by modulating signals from the suprachiasmatic nucleus, thereby potentially reducing delirium incidence. However, some studies have found no significant difference in delirium incidence compared with placebo, and robust evidence for its efficacy remains lacking. Another approach involves the use of antipsychotics such as haloperidol or olanzapine. Nevertheless, research indicates that haloperidol does not significantly shorten delirium duration and may be associated with higher six month mortality. High dose haloperidol can also induce cardiotoxicity, including QT interval prolongation, torsades de pointes, and hypotension. Additionally, GABA receptor agonists like benzodiazepines are used for sedation and anxiolysis in critically ill patients, yet prolonged use is believed to increase the risk of delirium. Dexmedetomidine, a potent and highly selective α 2 adrenergic receptor agonist, offers sedative, analgesic, anxiolytic, and opioid sparing properties. It is widely used in clinical practice and, compared with other sedatives, demonstrates advantages in reducing postoperative complications and shortening hospital length of stay. A prospective study in patients with type II respiratory failure receiving non intubated respiratory support compared dexmedetomidine, propofol, and remifentanil for sedation and analgesia. The dexmedetomidine group showed lower rates of non intubated respiratory support failure, lower mortality, and shorter ICU and hospital stays. However, no current guidelines recommend dexmedetomidine for managing agitation or delirium occurring during non intubated respiratory support.

Non intubated respiratory support is widely used in clinical practice, yet its failure rate is considerable. Studies report failure rates ranging from 15% to 38%-and up to 50% in some settings-among patients with acute respiratory failure. A proportion of these failures can be attributed to agitation or delirium during therapy. For example, one study found that 18.1% of ICU patients developed delirium during non intubated positive pressure ventilation, and delirium was independently associated with ventilatory failure. Poor tolerance due to anxiety or discomfort is considered a key driver of non intubated respiratory support failure. Another study reported an 18.18% incidence of delirium in patients receiving sequential high flow nasal cannula oxygen therapy after extubation. For cases of ventilatory failure secondary to agitation or delirium during non intubated support, moderate sedation is a recommended strategy to improve success rates. Although dexmedetomidine can reduce agitation duration in non intubated ICU patients, its effect on shortening delirium duration or preventing intubation remains uncertain, as suggested by the 4D trial in patients with hyperactive delirium. Moreover, dexmedetomidine significantly increases the risk of bradycardia and hypotension, and its labeling notes additional side effects such as headache, dry mouth, nausea, vomiting, and abnormal body temperature fluctuations.

Ketamine, a phencyclidine derivative, provides hemodynamically stable anesthesia through central sympathetic stimulation without significant respiratory depression. The combination of ketamine and dexmedetomidine has been associated with better mask or helmet compliance, faster sedation onset, and improved hemodynamic stability. Mechanistically, ketamine increases extracellular norepinephrine and dopamine concentrations in a time and dose dependent manner, whereas dexmedetomidine can cause bradycardia and vasodilation. Thus, their combination may produce counter balancing effects, yielding a net "negative negative positive" outcome. A multimodal regimen such as esketamine combined with dexmedetomidine for managing agitation or delirium during non intubated respiratory support could offer a promising approach to achieve rapid sedation, reduce delirium incidence, and maintain hemodynamic stability.

Esketamine, the S enantiomer of racemic ketamine, is considered approximately two to three times more potent than the racemate and is associated with a more favorable adverse effect profile, including fewer psychotomimetic symptoms. Low dose esketamine has been shown to reduce the incidence and severity of extubation related cough in patients undergoing laryngoscopic surgery and to decrease postoperative delirium incidence and pain levels in elderly surgical patients. In frail elderly patients undergoing laparoscopic radical resection for gastrointestinal tumors, low dose esketamine lowered delirium associated biomarker concentrations and effectively reduced postoperative delirium incidence. Currently, the combination of esketamine and dexmedetomidine has been employed in various settings, including intraoperative anesthesia, pediatric procedural sedation, gastrointestinal endoscopy, trauma analgesia, and mechanical ventilation. However, its utility for delirium occurring during non intubated respiratory support has not been formally evaluated. Our research group's earlier work confirmed that the combination is safe and effective for sedation in mechanically ventilated ICU patients, reducing ICU length of stay and time to awakening without increasing hypotension or bradycardia, compared with dexmedetomidine alone. Building on these preliminary findings, this study will investigate the efficacy and safety of esketamine combined with dexmedetomidine for the management of hyperactive delirium in ICU patients receiving non intubated respiratory support, with the aim of providing new insights to improve delirium related outcomes in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤90 years;
2. Hospitalized in the Intensive Care Unit (ICU) or receiving ICU-level care (with an expected ICU stay >24 hours);
3. Patients with hyperactive delirium: meeting criteria for CAM-ICU positivity (i.e., acute onset or fluctuating course plus inattention, and at least one secondary criterion-disorganized thinking or altered level of consciousness) and having a Richmond Agitation-Sedation Scale (RASS) score > +1. (The RASS and the Confusion Assessment Method for the ICU (CAM-ICU) are used to assess sedation and delirium levels. Hyperactive delirium is defined as CAM-ICU positive with RASS > +1);
4. Receiving non-intubated respiratory support (for >12 hours);
5. Body Mass Index (BMI) between 18 kg/m² and 30 kg/m² for each patient.

Exclusion Criteria:

1. Known or suspected allergy to any of the study drugs;
2. Acute myocardial infarction, severe arrhythmias (e.g., ventricular fibrillation, second- or third-degree atrioventricular block, sick sinus syndrome, ventricular tachycardia, QTc interval ≥470 ms, etc.), or left ventricular ejection fraction (LVEF) <30%;
3. Severe bradycardia (heart rate <40 beats per minute) with significant symptoms and hemodynamic instability;
4. Pregnancy or lactation;
5. Conditions that may affect efficacy assessment or cognitive function testing, such as blindness or deafness;
6. History of epilepsy or seizures;
7. Severe central nervous system disorders (e.g., cerebrovascular accident, coma, etc.);
8. Neuropsychiatric conditions per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) that may introduce bias (e.g., active substance use disorder, psychosis, etc.), including alcoholism, drug abuse, or use of psychotropic medications;
9. Patients receiving non-intubated respiratory support via a tracheostomy;
10. Patients with untreated or inadequately treated hyperthyroidism;
11. Patients with poorly controlled hypertension (resting systolic/diastolic blood pressure >180/100 mmHg);
12. Patients or their legally authorized representatives (family members) who are unable to cooperate or unwilling to provide written informed consent;
13. Severe hepatic insufficiency (Child-Pugh grade C);
14. Severe renal dysfunction, defined as: chronic renal insufficiency with a glomerular filtration rate (GFR) ≤ 29 mL/min/1.73 m²; or subjects on long-term maintenance hemodialysis or peritoneal dialysis;
15. A history of sleep disorders requiring medical intervention within the past month;
16. Other conditions deemed unsuitable for inclusion by the investigators.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-02-22 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Duration of Delirium (Time with positive CAM-ICU) | Usually within 30 days
  RASS assessments were performed at the 1st, 2nd, and 3rd hours (H1, H2, H3) after the administration of the study or control drug to randomized enrolled patients, followed by an assessment frequency of once every 2 hours thereafter, with scores recorded accordingly.
  If a patient who has become CAM-ICU negative and achieved an RASS score between -2 and +1 experiences a sudden recurrence of agitation or delirium, CAM-ICU and RASS assessments will be performed immediately and then repeated hourly until the patient is again CAM-ICU negative with an RASS between -2 and +1, or until non-invasive respiratory support is discontinued for any reason.

SECONDARY OUTCOMES:
Duration of Agitation (Time with RASS > +1) | Usually within 30 days
  After randomization, enrolled patients will be assessed using the RASS at hours 1, 2, and 3 (H1, H2, H3), followed by assessments every 2 hours, with all scores recorded.
Endotracheal Intubation and Mechanical Ventilation Rate | Usually within 30 days
  The rate of endotracheal intubation and mechanical ventilation during the study period will be calculated for each group (number of events / total number of patients in the group). The HACOR score will be assessed at enrollment (H0) and subsequently twice daily (between 08:00-10:00 and 16:00-18:00), with intervals exceeding 6 hours between assessments. All scores will be recorded.
28-day Mortality Rate | Usually within 30 days
  28-day all-cause mortality following study drug initiation
ROX Index and SpO₂/FiO₂ Ratio | Usually within 30 days
  After randomization, the ROX index and SpO₂/FiO₂ ratio will be calculated for enrolled patients at hours 1, 2, 3, 4, 5, and 6 (H1 to H6). Subsequently, these parameters will be assessed twice daily (between 08:00-10:00 and 16:00-18:00), with intervals exceeding 6 hours between assessments.
Length of ICU Stay | Usually within 30 days
  It is calculated from the time of ICU admission to the time of ICU discharge.
Incidence of Adverse Events | Usually within 30 days
  This includes electrocardiographic abnormalities (bradycardia, arrhythmia, myocardial ischemia, tachycardia, or QTc prolongation), hypotension or hypertension requiring any vasoactive medication, respiratory distress or apnea, and delirium-related complications (such as unplanned removal of catheters, tubes, or drains, increased secretions, etc.).
Use of Antipsychotic Medications | Usually within 30 days
  For patients whose agitation is not adequately controlled even after reaching the maximum dose of the study medication, haloperidol boluses may be administered every 10 to 30 minutes until agitation subsides (maximum total dose: 30 mg). The use of any other psychotropic medications will also be recorded.
Pain Assessment using the Critical-Care Pain Observation Tool (CPOT) or Visual Analog Scale (VAS) | Usually within 30 days
  Pain scores will be assessed at 15 minutes, 2 hours, 4 hours, and 24 hours after initiation of the study medication, and subsequently once every 24 hours.
Athens Insomnia Scale (AIS) Score | Usually within 30 days
  All enrolled patients will complete the AIS before receiving the study medication. The AIS will be administered again on the first morning after 24 hours of medication (at 10:00) and subsequently every morning (at 10:00), with all scores recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China